CLINICAL TRIAL: NCT07135557
Title: Evaluation of the Safety and Effectiveness of the R-One System in Percutaneous Coronary Interventions (PCI)
Brief Title: R-ONE® Robotically-Enhanced PCI Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cathbot (Shanghai) Robot Co., Ltd (Industry)
Collaborators: Chinese PLA General Hospital (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Shanxi Cardiovascular Hospital (Other); Meizhou People's Hospital (Other); Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CATHBOT-2021-R-One
Record Dates: First submitted 2022-11-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases
Keywords: PCI; Robotic; Cardiovascular
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The investigational device was R-One Vascular Interventional Navigation Control System and composed of following:
  The instruction unit is the control center and consists of a standby button, activation button, screen, acceleration button, stent/balloon catheter lever, guidewire lever, emergency stop button, guide rail, brake, and start/shutdown button.
  The robot consists of a table/support joint arm interface, table tilt button, fixture guide button, emergency stop button, release support arm brake button, and handles.
  The support joint arm consists of a support plate, a clamping clamp, a communication cable, a connector, and a support joint arm/table interface.
  The instruction unit protective sleeve consists of the operative field, the lever sleeve, and the shaper.
  The cartridge consists of cover, clamp backup, alternate path, guide path, wire guide slot, opening instruction of the rollers, and Y-connector clip.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evaluate safety and efficacy of the R-One vascular interventional navigation control system for PCI (Experimental)
  Interventions: Device: R-One vascular interventional navigation control system

INTERVENTIONS:
Device: R-One vascular interventional navigation control system — The interventional cardiologist sits at the cockpit and remotely performs the PCI using the console joysticks. The cassette, which is loaded with the interventional devices and connected to the guiding catheters, imposes axial and rotational forces on the intracoronary devices. Fluoroscopic, electrocardiographic, and hemodynamic images are "slaved" to the duplicate monitors inside the cockpit, enabling visualization from a closer distance. After completion of diagnostic angiography, the guiding catheter was positioned at the ostium of the coronary artery and connected to the disposable cassette on the robotic drive. The guidewire was loaded into the cassette. Treatment was administrated according to local site protocols. Pre and post dilation was done per operator discretion. All intracoronary devices were to be manipulated exclusively by the robotic system, with bailout to manual conversion when needed.

SUMMARY:
The aim of this study was to evaluate the safety as well as the clinical and technical effectiveness of robotic assisted percutaneous coronary intervention. This was a prospective, single-arm, multicenter, open-label, nonrandomized study. The study protocol was approved by the institutional review boards or local ethics committees of the participating facilities, and all patients provided written informed consent.

Patients with angiographic documentation of obstructive coronary artery disease and evidence of myocardial ischemia were enrolled in the study. Major inclusion criteria were stenosis of target vessel at least 50% by visual estimate, with maximal length of 34 mm and maximal diameter of 4.0 mm, that could be completely covered by a single stent. Major exclusion criteria included planned PCI or coronary artery bypass graft surgery, required treatment of more than 2 coronary artery or more than 1 lesion in each target artery, previous stent implantation within 5.0 mm of the target lesion, target lesion within 5 mm of the artery opening, planned treatment with directional or rotational atherectomy, intraluminal thrombus, severe tortuosity or calcification of the lesion or proximal to it, involvement of a bifurcation, or unprotected left main coronary artery.

All patients underwent PCI with the robotic R-OneTM System (R-One Vascular Robotics, Cathbot). The system was designed for coronary PCI and consists of 2 major components: the command unit and a bedside robot. The command unit is a radiation-shielded, mobile workstation that was positioned in the corner of the catheterization laboratory. The interventional cardiologist sits at the command unit and remotely performs the PCI using the console joysticks. Commands from the control console are delivered as electrical signals along a communication cable that runs from the control console to the robotic drive, on which a sterile cassette is placed. The cassette, which is loaded with the robot and connected to the guiding catheters, imposes axial and rotational forces on the intracoronary devices. The robotic-assisted system is compatible with all commercially available 0.014-inch guidewires, rapid-exchange coronary angioplasty balloons, and stent delivery systems. Fluoro-scopic, electrocardiographic, and hemodynamic images are "slaved" to the duplicate monitors inside the cockpit, enabling visualization from a closer distance. All operators had training on the system that included either animal laboratory experience or using the device to simulate operation before enrolling patients in the study.

After completion of diagnostic angiography, the guiding catheter was positioned at the ostium of the coronary artery and connected to the disposable cassette on the robotic drive. The guidewire was loaded into the cassette before starting the robotic-enhanced PCI. The treatment plan is decided by the doctor according to the patients' situation to perform pre-dilation, stent implantation, post-dilation, or drug balloon. All intracoronary devices were to be manipulated exclusively by the robotic system, with bailout to manual conversion when needed.

The primary endpoints were clinical procedural success and device technical success. Clinical procedural success was defined as <30% residual stenosis and Thrombolysis In Myocardial Infarction (TIMI) grade 3 at the completion of the procedure of robotically-treated lesions as determined by a quantitative coronary angiographic core laboratory, in the absence of major adverse cardiovascular events (MACE), either before hospital discharge or within 30 days of the procedure, whichever occurred first. Major adverse cardiovascular events were defined as cardiac death, Q-wave or non-Q-wave myocardial infarction, or clinically driven target vessel revascularization. All events were adjudicated by an independent clinical events committee. Device technical success was defined as the successful intracoronary advancement and retraction of the PCI devices (guidewire, balloon and stent) by the robotic system, without conversion to manual operation.

The necessary sample size for testing the endpoint of clinical and technical procedural success was calculated on the basis of the target value. The statistical analysis results show that the lower limit of the 95% confidence interval of the clinical success rate and the technical success rate of the operation is greater than 90% of the target value, and the invalid hypothesis is rejected. Both primary endpoints had to be met for the study to be declared successful. Data were analyzed on an intention-to-treat basis. Standard summary statistics were calculated for all patient and study outcome variables. Continuous variables were summarized using estimated means, standard deviations, minimums, maximums, medians, and interquartile ranges. Categorical data were summarized using frequencies, percentages, and 95% confidence interval.

DETAILED DESCRIPTION:
Purpose To evaluate the effectiveness of the R-OneTM vascular interventional navigation control system for percutaneous coronary interventions.

To evaluate the safety of the R-OneTM vascular interventional navigation control system for percutaneous coronary interventions.

Research design A prospective, multicenter, single-arm clinical trial. Subjects who met the inclusion criteria and did not meet the exclusion criteria were enrolled into the clinical study. The interventional cardiologists completed the robotic-assisted surgical operation using the investigational device during cardiovascular PCI treatment. The investigator is also required to evaluate the performance of the investigational device during the procedure and ultimately determine the safety and efficacy of its clinical application.

Device The investigational device was R-One Vascular Interventional Navigation Control System developed and produced by Robocath, and was composed of a platform (instruction unit, robot, support joint arm), a mobile radiation-proof screen, and a consumable set (cartridge, instruction unit protective sleeve).

Scope of Trial The subjects scope of the clinical trial: Patients requiring cardiovascular PCI.

Experimental Procedure Information of all the patients who have signed the Informed Consent Form and actually pass the screening will be registered in the screening/enrollment log sheet. If a subject is excluded from the trial, the investigator should specify the reasons for screening failure. If a subject is enrolled in the trial but does not use the investigational device, the reason should also be recorded.

All subjects enrolled in the trial will be given a corresponding enrollment number.

Introductory study population: The first 2 subjects enrolled at each clinical research center are considered to be the introductory study population. The introductory study population comply with the same protocol as the primary study population in follow-ups, but their results were analyzed separately and not included in the primary study population analysis Screening visit (baseline data collection) To collect the basic clinical information or complete relevant assessment in order to confirm whether the subject could be enrolled in the trial.

72-hour pre-operative collected ECG, cardiac enzyme, and concomitant medication records.

Operation day visit The investigator is also required to complete the cardiology robot-assisted surgical treatment using the investigational device and record the procedure, LED Scale, SME Scale, and device Performance Evaluation Pre-discharge visit The investigator shall collect the blood test, creatinine, ECG. cardiac enzyme, concomitant medication records.

1 month post-operative visit The investigator shall collect the concomitant medication records.

Application method of the investigational device Subjects who meet the inclusion criteria and do not meet the exclusion criteria will be enrolled in the clinical study and the interventional cardiologist will complete the therapeutic treatment on the subject while performing the cardiology PCI procedure.

The investigational devices should be used by investigators respectively during the surgical treatment according to product instructions . Interventional cardiologists who would participate in the trial and use the study device should have completed at least 80 PCI procedures and need to be trained and supervised by the physician who completed the animal experiments using the investigational device.

General procedure of a surgical operation

1. Connect the power cord to the mains.
2. Load the instruction unit, ensuring that the positioning mark on the base and that on the radiation-proof screen overlap.
3. Switch on the system
4. Activate the system.
5. Prepare R-One consumables kit.
6. Install the instruction unit protective sleeve.
7. Install the cartridge.
8. Install the robot.
9. Attach the Y-connector clip to the cartridge.
10. Insert the guide wire in the cartridge.
11. Navigate the guide wire through the instruction unit
12. Move the control lever and actuate the guidewire
13. Fix the guidewire
14. Insert the catheter into the cartridge
15. Navigate the catheter through the instruction unit
16. Move the control lever and actuate the catheter
17. Securing catheter
18. Simultaneous navigate the guidewire and catheter from the instruction unit
19. Place the guide wire in the alternate path as a backup
20. Place the catheter in the alternate path as a backup
21. Adjust the robot position

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

Subjects must meet all of the following inclusion criteria:

1. 18 years of age ≤ age ≤ 80 years of age.
2. Have clinical indication(s) for PCI and need to be treated with a PCI procedure.
3. Subjects voluntarily signed an informed consent form and were willing to complete follow-up visits.

Angiography Inclusion Criteria

1. Visual description of target lesion diameter stenosis ≥70% (or ≥50% accompanied with clinical evidence of myocardial ischemia within that range;
2. 2.5 mm ≤reference vessel diameter by visual description ≤ 4.0 mm.
3. Target lesion length ≤34.0 mm by visual description (If it is made up of multiple small lesions, the distance of which should not exceed 10 mm) and can be fully covered by a single stent. There are no less than 2.0 mm normal segmental vessels at the proximal and distal margins of the diseased region.
4. ≤2 target vessels to be treated, one single stent for each target lesion per target vessel, and target lesions can not be treated through stages.

Exclusion Criteria:

General Exclusion Criteria

Subjects cannot meet any of the following exclusion criteria:

1. Subjects have undergone other PCI within 72 hours prior to the R-One PCI procedure;
2. Subjects have undergone PCI within 30 days prior to the R-One PCI procedure and have experienced a MACE or other serious adverse event;
3. Acute myocardial infarction (MI) within one week prior to scheduled R-One PCI procedure;
4. Severe heart failure (NYHA ≥ Class III);
5. Cardiogenic shock within 48 hours prior to the PCI procedure;
6. Pregnant and lactating women, or women with plans to become pregnant during the clinical trial;
7. Subjects with allergies to aspirin, heparin, clopidogrel, contrast media, metallic materials and rapamycin;
8. Subjects with a platelet count <100 x 109/L or >700 x 109/L and a white blood cell (WBC) count <3 x 109/L (e.g., thrombocytopenia, thrombocytosis, neutropenia or leukopenia);
9. Subjects with creatinine levels ≥ 177 umol/L;
10. Subjects had a stroke within 30 days prior to the planned R-One PCI procedure.
11. Subjects with an active peptic ulcer or upper gastrointestinal hemorrhage within 6 months prior to the PCI procedure.
12. Subjects with a history of massive haemorrhage or coagulation disorder, or refusal of blood transfusion within the previous 6 months.
13. Subjects are currently enrolled in another clinical study that has not yet completed the entire follow-up period.
14. The investigators determined that the patient was not applicable for robot-assisted PCI.

Angiography Exclusion Criteria

1. TIMI blood flow grade of <3 for the target lesion.
2. In-stent restenosis, or the target vessel has implanted a stent previous which in close proximity to the target lesion.
3. Need other treatments (e.g., atherectomy or laser treatment) in addition to balloon angioplasty and stentoplasty.
4. 2 or more lesions in a single vessel that need treatment concurrently;
5. Bifurcation lesions requiring protection;
6. Visible thrombosis;
7. Target lesion located in the left coronary artery trunk;
8. Target lesion within 5 mm of left anterior descending (LAD), left circumflex (LCX) or right coronary artery (RCA) opening;
9. Severe distorted and/or calcified lesions, and its coronary anatomy is not applicable for robot-assisted PCI according to the the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Clinical success rate of the surgery | Day of surgery
  Clinical success rate = number of subjects that were clinical successes ÷ number of subjects that received surgical treatment × 100%.
  Evaluation Method:
  1. The target lesion was treated with test device, and the residual stenosis in the target vessel (visual description by angiography) reduced to less than 30% after PCI and a TIMI grade of 3.
  2. No major adverse cardiovascular events (MACE) occurred in the hospital.
Success rate of surgical techniques | Day of surgery
  Technical success rate = number of subjects that were technical successes ÷ number of subjects received surgical treatment × 100%
  Evaluation Method:
  The Robot-assisted PCI procedure was successfully completed without any unplanned manual assistance or shift to manual operation.
  1. Definition of planned manual assistance:
     During robotic surgery: Reposition of guidewires or stents/balloons, manual translation/rotation of guidewires or stents/balloons to guiding catheters, reposition of guiding catheters and usage of any device that is not compatible with the robotic platform
  2. Definition of unplanned manual assistance:
     Manual translation/rotation of the guidewire and/or manual translation of the stent/balloon once the guidewire has left the guiding catheter
  3. Definition of the shift to manual operation:
  Any situation during the PCI procedure that results in the shift to manual operation.
  System restart failure during robotic surgery

SECONDARY OUTCOMES:
Procedure duration | Day of surgery
  Procedure duration = arterial sheath removal time - arterial sheath insertion time
Duration of robot-assisted treatment | Day of surgery
  Robot-assisted treatment duration = time when the robot finish moving the guidewire away from the coronary vessel - time when the robot start to move the guidewire away from the guiding catheter
Radiation exposure to the patient | Day of surgery
  Evaluation Method: Measure and record dose exposure by angiography (DSA)
Radiation exposure to interventional cardiologists | Day of surgery
  Detect radiation through radiation dosimeters. Two dosimeters will be used simultaneously during the procedure. One is placed on the operating table and the other is worn by the interventional cardiologist to measure the radiation dose exposed to the interventional cardiologist. Both dosimeters will be calibrated once a day before use and reset to zero before each PCI procedure. Radiation readings from the dosimeter will be recorded when the first guidewire is inserted into the vessel and the last guidewire is pulled out of the vessel.
Contrast dose | Day of surgery
  Record the contrast dose used during intra-operative angiography
MACE | Day of surgery and 1 month post-operative
  Record the in-hospital MACE of subjects Record the MACE occurred 1 month (30±7 days) after the PCI procedure

OTHER OUTCOMES:
Evaluate intra-operative physiological load of interventional cardiologists | Day of surgery
  Interventional cardiologists are required to complete the Local Experienced Discomfort Questionnaire (LED scale) in time after the surgery in order to provide a retrospective evaluation of the physiological sensations during the procedure in the way of visual analog scale.0 = No discomfort at all, and 10 = Very uncomfortable.
Intraoperative psychological load evaluation of interventional cardiologists | Day of surgery
  Interventional cardiologists are required to complete the Subjective Mental Effort Questionnaire (SME scale) in time after the surgery in order to provide a retrospective evaluation of the mental feelings during the procedure in the way of visual analog scale. 0 = Not difficult at all, and 100 = Extremely difficult.
Incidence rate of serious system malfunction | Day of surgery
  Incidence rate of serious system malfunction = Number of procedures with serious system malfunction during robot-assisted surgery ÷ Number of procedures in which robot-assisted surgery was performed × 100%.
  Evaluation Method:
  Definition of serious system malfunction: System malfunctions that occur during robot-assisted surgery that are difficult to repair in a short period of time and can have a serious impact on the surgical process or options.
The occurrences of repairable system malfunction | Day of surgery
  Definition of repairable system malfunction: Simple malfunctions that occur during robot-assisted surgery that can be repaired by a technician or the surgical team and do not have a serious impact on the surgical process or options.
Evaluation of Device Usability | Day of surgery
  Investigators are required to complete the Device Performance Record after surgery and provide a retrospectively evaluation of performance of the investigational device during the trial, with the grades from high to low being excellent, good, medium, and poor.
Indicators for Safety Evaluation | 72 hours pre, day of surgery, from the postoperative period to discharge (average discharge 3-5 days after surgery, the maximum follow-up period shall not exceed one month), 1-month post-operative add or subtract 7 days
  Subjects' laboratory test results of blood routine, myocardial enzymes, creatinine, etc. during the screening period, operation day, pre-discharge and 1-month post-operative visit. The results were reported according to the reference range (normal/abnormal and meaningful/abnormal and not meaningful).
The occurrences of of Adverse Events | Day of surgery, from the postoperative period to discharge (average discharge 3-5 days after surgery. If discharge is delayed due to PCI complications, the maximum follow-up period shall not exceed 1 month), 1-month post-operative add or subtract 7 days
  Record and report all information of adverse events during the clinical trial, as well as investigational device-related adverse events and serious adverse events.
  Definition of adverse events: Adverse events that may result from PCI surgery and anesthesia include angina pectoris, myocardial infarction, myocardial infarction recurrence, acute coronary artery occlusion, no-reflux, coronary artery perforation, in-stent thrombosis, stent dislodgement, haemorrhage, vascular complications, contrast-induced acute kidney injury, MACE, adverse reactions to anesthesia, allergic reaction, death.
  Definition of serious adverse events: death, life-threatening, hospitalization required or prolonged hospitalization, disability, affect the ability to work, or cause congenital deformities, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, Principal Investigator — Chinese PLA General Hospital
Locations (4):
- China (4):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No